CLINICAL TRIAL: NCT01644305
Title: 1. Association of Plasma GDF-9 or GDF-15 Levels With Bone Parameters in Polycystic Ovary Syndrome. 2. Plasma GDF-15 Levels and Their Association With Hormonal and Metabolic Status in Women With Polycystic Ovary Syndrome Aged 25-35.
Brief Title: Plasma Levels of GDF-9 and GDF-15 in Patients With Polycystic Ovary Syndrome.
Status: Completed | Type: Observational
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zehra Berberoglu, Ass. Prof., Ankara Education and Research Hospital
Other Study IDs: 3849
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Polycystic Ovary Syndrome
- Idiopathic hirsutism
- Control

SUMMARY:
The purpose of this study is to determine the plasma levels of GDF-9 and GDF-15, and their association with bone and cardiovascular parameters in patients with Polycystic Ovary Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Female patients at ages 25-35 diagnosed with polycystic ovarian syndrome and idiopathic hirsutism

Exclusion Criteria:

* acute infectious disease, a thyroid, pituitary, nutritional, inflammatory, hepatic, renal, or neoplastic disorder; history of cardiovascular disease or pulmonary embolism; a family history of coronary artery disease; smoking history; hypertension; diabetes mellitus; use of oral contraceptives, anti-androgens and drugs known to interfere with cytokine release, such as corticosteroids, immunosuppressors, or nonsteroidal antiinflammatory drugs.

any medication known to affect hormonal or metabolic parameters.

Ages: 25 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Hospital Endocrinology Outpatient Clinic
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
The association of GDF 9 AND GDF 15 with bone and cardiovascular parameters in women with polycystic ovary syndrome | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Education and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berberoglu Z, Aktas A, Fidan Y, Yazici AC, Aral Y. Association of plasma GDF-9 or GDF-15 levels with bone parameters in polycystic ovary syndrome. J Bone Miner Metab. 2015 Jan;33(1):101-8. doi: 10.1007/s00774-013-0560-8. Epub 2014 Jan 16. PMID 24430093